CLINICAL TRIAL: NCT02474030
Title: Relationship Between Electrical Pain Tolerance Threshold of Alveolar Ridge and Individual Attributes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nihon University (Other)
Responsible Party: Principal Investigator, Yoshio Nakashima, Department of Removable Prothodontics, Nihon University
Other Study IDs: EC 13-12-003-3
Record Dates: First submitted 2015-06-11; First posted 2015-06-17 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Intraoral Pain Threshold

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This study was conducted with an aim to know how individual attributes associated to intraoral Pain Tolerance Threshold. The hypotheses were that the Pain Tolerance Threshold associated to age, sex, prosthodontic oral condition evaluated by the Eichner Index, and psychological state evaluated by the Profile of Mood States.

ELIGIBILITY:
Inclusion Criteria:

* not pacemaker wearers

Exclusion Criteria:

* general health problems that could affect the measurement of nerve activity a lack of understanding of written or spoken Japanese

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers participants studying or workung at the Nihon University School of Dentistry at Matsudo took part in the study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
pain threshold | 20minutes
  intraoral electrical pain threshold

CONTACTS AND LOCATIONS:
Locations (1):
- Nihon University School of Dentistry at Matsudo, Matsudo, Chiba, Japan